CLINICAL TRIAL: NCT06364735
Title: Entities and Variables Related to Catch-up Growth in Pediatric Patients With Celiac Disease (CD) on a Gluten-free Diet (GFD)
Brief Title: Entities and Variables Related to Catch-up Growth
Status: Recruiting | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Elena Groppali, MD, ASST Fatebenefratelli Sacco
Other Study IDs: Entità e variabili
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Celiac Disease in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective monocentric observational no-profit study with the aim of evaluating the entity and potential variables influencing the catch-up growth of childhood gluten-free diet patients with celiac disease during a 10-year follow-up. The only extrapolation of the data collected in anonymized form from the medical records of patients who match the necessary study criteria will be planned in order to achieve this aim. A 900-patient sample size will be planned.

ELIGIBILITY:
Inclusion Criteria:

* celiac disease diagnosis established at the V. Buzzi Children's Hospital in Milan between January 2010 and December 2020, excluding the extremes, in accordance with the ESPGHAN 2012 or 2020 recommendations.

Exclusion Criteria:

* patients with unclear or non-specific duodenal histological alterations (e.g., atrophy with unavailable or negative specific antibodies for celiac disease);
* patients with additional chronic illnesses;
* absence of the data required for the study;
* patients with IgA deficiency, defined as IgA <20 mg/dl in children <3 years old or with levels that are below normal for their age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Childhood celiac disease patients on a gluten-free diet
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Measure the catch-up growth degree. | 6 and 24 month
  Changes in the auxological weight variable in pediatric patients with celiac disease were measured 6 months and 24 months after they started a gluten-free diet. The change was expressed as an average daily weight increase and compared with the average increase expected for sex and age in a healthy population extrapolated from validated curves (Cacciari).

SECONDARY OUTCOMES:
Calculate the degree of catch-up growth | 6 and 24 month
  Variation in the auxological variable of height in pediatric patients with celiac disease, measured as variation in the standard deviation of this variable compared to reference values for age and sex extrapolated from validated curves (Cacciari curves), at six and twenty-four months after the start of the gluten-free diet.

OTHER OUTCOMES:
Exploratory objectives 1 | 6 and 24 month
  Identify the correlation between the degree of catch-up growth and the persistence of the symptoms, MC-related antibody positivity and the level of diet adherence at the 6- and 24-month follow-up
Exploratory objectives 2 | 6 and 24 month
  Define the degree of celiac disease's clinical, endoscopic, histological, and serological severity at the time the sample was diagnosed, and then correlate it to the degree of catch-up growth that occurred 6 and 24 months after the gluten-free diet was started

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No